CLINICAL TRIAL: NCT06438250
Title: 68Ga-JH04 PET/CT: Dosimetry and Biodistribution Study in Patients With Various Cancers
Brief Title: 68Ga-JH04 PET/CT: Dosimetry and Biodistribution Studies
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FirstAHFujian-68Ga-JH04
Record Dates: First submitted 2024-05-27; First posted 2024-05-31 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Drug: 68Ga-JH04
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- dynamic PET scans (Experimental): PET imaging will begin at 3 minutes, 15 minutes, 30min minutes, 60 minutes and 150 minutes after injection
  Interventions: Drug: 68Ga-JH04

INTERVENTIONS:
Drug: 68Ga-JH04 — The dose will be 148-222 MBq given intravenously.

SUMMARY:
68Ga-JH04 is a novel radiotracer targeting fibroblast activation protein (FAP). In this study, we observed the safety, biodistribution, and radiation dosimetry of 68Ga-JH04 in patients with different types of cancer.

DETAILED DESCRIPTION:
Carcinoma-associated fibroblasts (CAFs) are an integral part of the tumor microenvironment, and fibroblast activation protein (FAP), as a specific marker of CAFs, is overexpressed in more than 90% of epithelial malignant tumors' CAFs, with limited expression in normal tissues, making it an appropriate target for various tumors. Currently, several tracers targeting FAP for diagnostic purposes have been developed, such as 68Ga-FAPI-04, 68Ga-FAPI-02, and showed high efficacy in tumor staging and restaging. 68Ga-JH04, a novel radiopharmaceutical targeting FAP, demostrated high stability in vitro and in vivo, and can accumulate specifically in tumors with high binding affinity, safety, and selectivity in preclinical studies. In this study, the safety, biodistribution, and radiation dosimetry of 68Ga-JH04 in patients with different types of cancer were observed to evaluate the dosimetric characteristics of 68Ga-JH04.

ELIGIBILITY:
Inclusion Criteria:

* Various solid tumors with available histopathological findings
* Signed informed consent

Exclusion Criteria:

* pregnant or lactational women
* who suffered from severe hepatic and renal insufficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
safety and tolerability | Up to 1 week
  Hematologic status, liver function, renal function and General vital signs were recorded before and 1 week after administration of radiopharmaceutical. Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
Human biodistribution | From right after tracer injection to 150 minutes at post-injection
  reported as relative uptake values per organ at 3 minutes, 15 minutes, 30 minutes, 60 minutes and 150 minutes per individual subject and as a mean over all subjects
Human dosimetry | From right after tracer injection to 150 minutes at post-injection
  radiation dose to individual organs and the equivalent dose for the whole body of each subject and as a mean over all subjects. Dosimetry will be calculated using the Hybrid-Dosimetry software.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — The First Affiliated Hospital, Fujian Medical University
Locations (1):
- Department of Nuclear Medicine, First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No